CLINICAL TRIAL: NCT01182662
Title: Phase II Study of Umbilical Cord/Placenta-Derived Mesenchymal Stem Cells to Treat SAA
Brief Title: Safety and Efficacy Study of Umbilical Cord/Placenta-Derived Mesenchymal Stem Cells to Treat Severe Aplastic Anemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Chengyun Zheng, Department of Hematology of the 2nd Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kongdx; No. 30670903 (Other: National Natural Science Foundation of China)
Record Dates: First submitted 2010-08-11; First posted 2010-08-17 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Aplastic Anemia
Keywords: Bone Marrow Disease; Aplastic Anemia; Umbilical Cord/placenta-Derived MSC; Transplantation
MeSH Terms: conditions — Anemia, Aplastic; Bone Marrow Diseases | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human umbilical cord-derived MSCs and cyclosporin (Experimental): Human umbilical cord-derived MSCs at a dose of 1.0E+6 MSC/kg, repeated to apply in trimonthly for 2 cycle and CsA 5mg/kg po for 12 months
  Interventions: Other: Human umbilical cord-derived MSCs and cyclosporin A
- cyclosporine A (Active Comparator): cyclosporine A at a dose of 5 mg CsA/kg
  Interventions: Other: cyclosporin A

INTERVENTIONS:
Other: Human umbilical cord-derived MSCs and cyclosporin A — 1.0E+6 MSC/kg, IV drop and repeat to apply in trimonthly for 2 cycle and cyclosporin A 5mg/kg po for 12 months
  Arms: Human umbilical cord-derived MSCs and cyclosporin
Other: cyclosporin A — cyclosporin A 5mg/kg po for 12 months
  Arms: cyclosporine A

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mesenchymal stem cells (MSCs) derived from human umbilical cord/placenta at a dose of 1.0E+6 MSC/kg in subject for the therapy of severe aplastic anemia (SAA).

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a condition that involves a low level of red blood cells, white blood cells, and platelets without evidence of another bone marrow disease. Patients with severe aplastic anemia produce too few blood cells, causing fatigue, easy bruising and bleeding, and susceptibility to infections. In many cases, the very low blood counts result from an autoimmune process. The patient's own immune system damages their stem cells in bone marrow.

Although immune-suppressing drugs, such as corticosteroids, CsA and ATG, have been used in the treatment of SAA, however, many studies have indicated that the overall response rate to these drugs is less than 60%. Addition, the severe side effects of these immune-suppressing drugs have also been observed. The management of SAA patients therefore remains unsatisfactory and targeted therapies are needed. Human MSCs isolated from human umbilical cord/placenta have been shown to have immunosuppressive, stimulating hematopoiesis and tissue repairing properties. This study will evaluate the safety and effectiveness of MSC transplantation in the SAA patients.

This study will last 2 to 3 years. Participants will be randomly assigned to receive either MSC transplant and CsA therapy (experimental group) or CsA therapy alone (control group). Patients will undergo MSC transplant at the start of the study on Day 0. After 3 months, patients will receive the second MSC transplantation. After six and twelve months from the first transplantation, patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18~80 years old with plan to infuse MSCs.
2. Standard of diagnosis of aplastic anemia is according to Chinese domestic classification of AA for 1987.
3. Patients must have an ECOG 0~2.
4. No moderate or sever organ dysfunction: Ejection fraction>45%; Creatinine <176 umol/L.
5. No active severe viral or fungus infection.
6. Each patient must sign written informed consent.

Exclusion Criteria:

1. Psychiatric condition that would limit informed consent.
2. HIV positive
3. Positive Pregnancy Test
4. Patient has enrolled another clinical trial study within last 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
SAA clinical symptoms | 1 year
  Anemia symptoms, bleeding and infection will be mainly observed in every monthly after transplanting MSCs for one year.
The number of blood cells | 1 year
  The number of blood cells, which contains WBC, Neu, RBC, Hb,PLT and reticulocyte, will be mainly tested monthly after transplantion of MSCs for one year
Bone borrow hemocytology | 1 year
  Bone borrow cytomorphologic examination will be tested in every 3 months after transplantion of MSCs for one year.

SECONDARY OUTCOMES:
Percentage of systemic T regulatory cell population and T lymphocyte subsets | 1 year
  Percentages of T regulatory cell population and T lymphocyte subsets in peripheral blood will be tested in every 3 months after transplanting MSCs for one year.

CONTACTS AND LOCATIONS:
Overall Officials: chengyun zheng, Ph. D, Principal Investigator — Department of Hematology of The 2nd Hospital of Shandong University
Locations (1):
- Department of Hematology of the 2nd Hospital of Shandong University, Jinan, Shandong, China